CLINICAL TRIAL: NCT01604616
Title: Short Term Postoperative Tamponade Using Perfluorocarbon Liquid for Giant Retinal Tears
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0032-12-ZIV
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Retinal Detachment
MeSH Terms: conditions — Retinal Detachment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- PCFL GROUP: patients in this group had the PFCL for a period of 7-10 days before it was replaced by SF6 gas or silicone oil
- control group: in thos group no PFCL was left in the eye and either SF6 or silicone oil was the definitive treatment at the time of the retinal detachment surgery repair.

SUMMARY:
The purpose of the article is, to investigate the efficacy and safety of perfluorocarbon liquid (PFCL) ,as a short term postoperative tamponade for treating retinal detachment ,associated with giant retinal tears.

DETAILED DESCRIPTION:
a retrospective study wich compared 2 groups that had giant tear repair in one group, PFCL was left for few days as an intermediate measure until silicone oil or SF6 gas was used to reattach the retina ,and in the control group SF6 or Silicone oil were used, with no PFCL.

ELIGIBILITY:
Inclusion Criteria:

* above 18 years of age
* retinal tear at least of 3 clock hours.

Exclusion Criteria:

* less than 18 years of age
* Retinal tear less than 3 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: man and women above the age of 18 years
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 1998-01; Study Completion 2012-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph pikkel, M.D, Principal Investigator — Ziv Medical Center
Locations (1):
- Ziv Medical Center, Safed, Israel